CLINICAL TRIAL: NCT00668798
Title: Incidence and Clinical Outcome of Human Cytomegalovirus Transmission Via Thawed Frozen Breast Milk in Preterm Infants <31 Weeks. A Prospective Trial.
Brief Title: Cytomegalovirus (CMV) Transmission by Frozen Breast Milk in Preterms
Status: Suspended | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof Karl Bauer, Head of Dpt. of Neonatology, Goethe University, Frankfurt
Other Study IDs: CMV/MM0105/FFM
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2008-04-29 (Estimated); Status verified 2008-04

CONDITIONS: Cytomegalovirus
Keywords: cytomegalovirus breast milk preterm infants transmission; transmission of CMV via thawed frozen breast milk

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — thawed frozen breast milk of lactating mothers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: mother CMV positive
- B: mother CMV negative

SUMMARY:
Cytomegalovirus infection threatens preterm infant. We investigated, whether thawed breast milk is a mode of transmission

DETAILED DESCRIPTION:
Preterm infants are at risk of symptomatic human cytomegalovirus infections transmitted by breast milk. This study evaluates incidence, timing, and clinical rlevance of acquired human CMV infections in preterm infants younger than 32 weeks of gestational age receiving maternal thawed frozen breast milk until 33 completed weeks of gestational age.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants of less than 32 weeks of gestation

Exclusion Criteria:

* preterm infant of 32 weeks of gestational age or older, feeding with solely formula milk
* ourborn infants
* retroviral infection
* CMV status of mother unclear
* informed consent missing

Ages: 24 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm infants of less than 32 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Estimated); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
CMV status of preterm infants | 2005-2008

SECONDARY OUTCOMES:
clinical manifestations of CMV infection | 2005-2008

CONTACTS AND LOCATIONS:
Overall Officials: Karl Bauer, Professor, Principal Investigator — Goethe University, Dpt of Neonatology
Locations (1):
- Childrens Hospital Goethe University, Frankfurt, Germany

REFERENCES:
- [Background] Hamprecht K, Maschmann J, Vochem M, Dietz K, Speer CP, Jahn G. Epidemiology of transmission of cytomegalovirus from mother to preterm infant by breastfeeding. Lancet. 2001 Feb 17;357(9255):513-8. doi: 10.1016/S0140-6736(00)04043-5. PMID 11229670